CLINICAL TRIAL: NCT00479960
Title: Effect of Dietary Supplementation With Omega-3 Fatty Acids on Human Sperm Characteristics, a Preliminary Study
Brief Title: A Preliminary Study on Effect of Omega-3 on Human Sperm
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Shaare Zedek Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 022006
Record Dates: First submitted 2007-05-28; First posted 2007-05-30 (Estimated); Last update posted 2007-05-30 (Estimated); Status verified 2006-11

CONDITIONS: Oligospermia
Keywords: Asthenozoospermia; Azoospermia; Oligospermia; Omega-3; Fatty Acids
MeSH Terms: conditions — Oligospermia; Asthenozoospermia; Azoospermia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: commercially available omega-3 fatty acids supplementation

SUMMARY:
The phospholipids of mammalian spermatozoa possess a distinctive fatty acid composition with high proportion of long chain polyunsaturated fatty acids. The lipid composition is a major determinant of the membrane flexibility and sperm motility required for proper fertilization. It also influences the sperm plasma membrane's fluidity, chilling sensitivity and thermotropic lipid phase transition (LPT) and these parameters determine our ability to cryopreserve these cells. Our hypotheses is that by providing dietary supplementation of omega-3 polyunsaturated fatty acids an improvement of sperm parameters (number, motility, viability) can be achieved. We also expect alteration spermatozoal plasma membrane fatty acid composition, making it more chilling resistant.

Experimental methodology: 1) Characterize fatty acid composition of the spermatozoa of normal and abnormal spermatozoa by gas chromatography. 2) Characterize sperm plasma membrane LPT by FTIR spectrometer. 3) Run a randomized double-blind, placebo controlled, crossed-over dietary fatty acid supplementation pilot trial in human sub-fertile patients. Large scale trial will follow, if justified. In both trials sperm characterization of each participant will be conducted before, during and following the trial.

Subfertile males will benefit greatly if their sperm parameters can be improved and cryopreserved while ensuring enhanced post-thawing survival. We believe that changing the fatty acid composition of sperm plasma membrane by simple dietary means will open the way to improve the fertility of those that needs it the most.

DETAILED DESCRIPTION:
The phospholipids of mammalian spermatozoa possess a distinctive and highly unusual fatty acid composition, the most unique feature of which is a very high proportion of long chain (C20-22) highly polyunsaturated fatty acyl groups. In most mammals, docosahexaenoic acid (DHA; 22:6,n-3) is the dominant polyunsaturated fatty acid (PUFA) although, in several species, docosapentaenoic acid (22:5,n-6) is also a major component 2. The lipid composition is a major determinant of the membrane flexibility required for the characteristic flagella movement of spermatozoa and for the fusogenic properties of the membranes associated with the acrosome reaction and fertilization. In addition, it has been demonstrated that lipid-derived mediators are involved in various signal transduction mechanisms that regulate spermatozoa functions.

Sperm motility was therefore closely correlated with fertility, yet factors controlling sperm motility in humans are not fully understood 12. The amount of PUFA, mainly DHA, and to a lesser extent eicosapentaenoic acid (EPA), was showed to be positively associated with sperm motility and essential for optimal fertility. The reduction in the amount of DHA in sperm lipids have been correlated with reduced sperm concentration, sperm progressive motility and the proportion of cells with normal morphology. In asthenozoospermic (poor sperm forward motility), the levels of DHA (and total PUFA) was found to be lower than in normozoospermic individuals despite similar serum fatty acid composition 18. Broiler spermatozoa rich in EPA or DHA or both showed significantly increased fertility following artificial insemination (AI).

Chilling injury to mammalian gametes has been described as the irreversible damage that occurs upon cooling to low, but non-freezing, temperatures. Several studies suggested that chilling injury is the major limiting factor for successful gamete cryopreservation. Other studies suggested that membranes are the primary sites for structural and functional chilling injury in sperm and oocytes. Additionally, membrane chilling injury is dependent on the biochemical and biophysical properties of membranes. The plasma membrane thermotropic lipid phase transition (Tm) from the fluid liquid crystalline phase to the more rigid gel phase is associated with chilling injury. When membrane lipids undergo lipid phase transition (LPT), fluidity decreases and the structure and functioning of the membrane change. As a result, the membrane permeability increases and the cells are damaged. The temperature at which Tm occurs is greatly affected by the fatty acid composition of the membrane. Membranes consisted of lipids with multiple unsaturations or short carbon chains are more fluid at low temperatures. The ability of the spermatozoal plasma membrane to resist structural damage during cryopreservation may therefore be related to its fatty acids composition and the strength of the bonds between membrane components 38. It was shown, for example, that spermatozoa of Asian elephants, which are more chilling sensitive than African elephant sperm, contain lower concentration of PUFA in their membranes and are especially poor in DHA.

There are several ways to change the chilling sensitivity and Tm in mammalian gametes. Spermatozoa can spontaneously interact with liposomes as was described in several studies. Previous work suggested that phospholipids adsorbed on to the sperm cells, which were then cooled to 4oC, increased the chilling resistance of the sperm cells from bovine, ram and elephant.

The relationship between dietary components and reproduction is well established. Follicular maturation, ovulation and oestrus in the female, and libido and fertility in the male, might all be adversely affected by undernutrition. Men with infertile semen were found to consume less omega-3 fatty acids than fertile men, and a significant correlation was established between the consumption of alpha-linolenic acid (18:3n-3) on the one hand and sperm concentration and progressive motility on the other hand. In boar, the output of the accessory glands, but not the output of spermatozoa by the testes, was affected by the reduced feed intake and is likely to reflect a suppression of androgen secretion. Various reports showed that enrichment of diet with PUFA can alter the biophysical properties or reproductive performance of mammalian and avian sperm and oocytes.

Objectives and expected significance of the research Male patients arriving at the male fertility clinic frequently suffer from one or more of the following: asthenozoospermia (low progressive motility), teratozoopermia (abnormal morphology) and/or oligozoospermia (low sperm count), collectively known as O.T.A It is assumed that by supplementing the diet of such patients with omega-3 PUFA, an improvement of these parameters can be achieved. Since the number of normal cells in all such patients is limited, omega-3 PUFA supplementation may confer the needed change to the sperm plasma membrane, making these cells more resistant to chilling injury during preservation. This will provide us with a mean to ascertain that more of the normal cells will survive the freezing and thawing processes involved in cryopreservation. By achieving that we will be able to make sure that enough normal cells will be available for fertilization.

If the hypothesis of this study is proved correct, it will mean that by a simple dietary mean we will be able to improve reproduction in those that needs it the most.

Comprehensive description of the methodology and plan of operation

1. Experimental design: The experiment will be a randomized double-blind, placebo controlled, crossed-over trial. The experiment will start with a pilot which will be conducted on 20 participants, all of which are out-patients at the male fertility clinic of the Shaare Zedek Medical Center, Jerusalem, Israel. The pilot is expected to be followed by a large scale trial in a similar design (without the "cross-over" part). Both pilot and large scale trial will seek and obtain the approval of the Helsinki committee of the Shaare Zedek Medical Center prior to their initiation. All participants will be asked to sign an informed consent.
2. Basic spermatozoa database: For general information on human spermatozoa, fresh and frozen samples of normal and subfertile males will be analyzed for total lipids fatty acids composition by gas chromatography. All samples will be evaluated for basic sperm quality characteristics according to the World Health Organization (WHO) guidelines 66. Samples will then be separated from the seminal plasma and stored till fatty acid composition analysis. Determination of the lipid phase transition temperatures by the FTIR spectrometer on fresh samples will also be conducted.
3. Dietary supplementation: At the beginning of the trial each participant will be provided with 120 capsules of either placebo or commercially available omega-3 fatty acids. The capsules will be consumed in the following manner: 2 capsules daily during the first week, 3 capsules per day during the second week and starting on the third week, 4 capsules per day till all are consumed. At this point there will be a break of 4 weeks before switching between the groups and resuming the same protocol once again. During the entire period each participant will also be provided with vitamin E pills as anti-oxidant.
4. During and post-experimental sperm characterization: Each of the participating patients will provide 5 samples during the dietary supplementation pilot experiment: Once at the beginning of the trial, once in the middle of each of the two segments (see dietary supplementation paragraph for details), once at the cross-over point and once at the end of the trial. All samples will be analyzed in the same way as described above.
5. Lipid phase transition determination: Approximately 10 of the participants in the pilot trial will be requested to provide additional samples at the cross over point and at the end of the trial for the determination of the lipid phase transition temperatures by the FTIR spectrometer. These participants will be selected based on their sperm fatty acid composition at the beginning of the trial so as to cover as wide range of compositions as possible.
6. Large scale trial: After analyzing the results of the pilot trial, a decision will be made if there is indication to proceed with a large scale trial. Assuming the results will indicate such a need, a large scale trial will be conducted. Experimental design will be randomized double-blind, placebo-controlled trial. The number of participating patients will be determined at the time the decision to proceed with such a trial will be made. At that time a decision will also be made what other male fertility clinics from additional medical centers to invite to participate.

ELIGIBILITY:
Inclusion Criteria:

* Patients with asthenozoospermia (low progressive motility), teratozoopermia (abnormal morphology) and/or oligozoospermia (low sperm count)

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2007-06; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
sperm count | 10 weeks

SECONDARY OUTCOMES:
sperm Lipid phase transition determination | 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Revel, MD, Principal Investigator — Hadassah university hospital
Locations (1):
- Shaare Zedek Medical Center, Jerusalem, Israel